CLINICAL TRIAL: NCT00991172
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Subcutaneously Administered REGN475 in Patients With Sciatic Pain
Brief Title: A Study to Evaluate the Safety and Efficacy of Subcutaneously Administered REGN475(SAR164877) in Patients With Sciatic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R475-PN-0908
Record Dates: First submitted 2009-09-04; First posted 2009-10-07 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Sciatica
Keywords: sciatica; sciatic pain; pain; back pain
MeSH Terms: conditions — Sciatica; Pain; Back Pain | interventions — fasinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo injection (Placebo Comparator)
  Interventions: Drug: Placebo Injection
- active (Experimental): subcutaneous injection of REGN475
  Interventions: Drug: REGN475
- active 2 (Experimental): subcutaneous injection of REGN475
  Interventions: Drug: REGN475

INTERVENTIONS:
Drug: REGN475 — Single Subcutaneous injection dose level 1
  Arms: active
Drug: REGN475 — Single subcutaneous injection dose level 2
  Arms: active 2
Drug: Placebo Injection — Placebo Subcutaneous injection
  Arms: placebo injection

SUMMARY:
This is a phase 2, randomized, double-blind, parallel-group, single dose study to evaluate the safety and efficacy of 2 dose levels of REGN475 compared with placebo in patients with sciatic pain. Enrollment of approximately 50 patients in each of the 3 treatment arms is expected at up to 35 US sites, for a total enrollment of approximately 150 patients. Patients will receive 1 injection under the skin of either active or placebo REGN475, and be followed over 10 visits for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Pain present for at least 2 weeks, but not lasting for more than 16 weeks prior to the screening visit.
2. A confirmed diagnosis of sciatica at the screening visit.
3. Weight less than 120 kg

Exclusion Criteria:

1. Back surgery within 6 months prior to the screening visit
2. Neurological deficit (muscle weakness and/or reflex loss; loss of bowel or bladder function) from any cause including sciatica
3. Other conditions which may confound the interpretation of the study, such as carpal tunnel syndrome, MS, rheumatoid arthritis, spinal stenosis, etc.
4. Allergy to doxycycline or related compounds
5. Women who are pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Sciatic pain between baseline and end of week 4 | 4 weeks

SECONDARY OUTCOMES:
Additional measures of sciatic pain. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tiseo, PhD, Study Director — Regeneron Pharmaceuticals
Locations (30):
- United States (30):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Mobile, Alabama
  - Regeneron Investigational Site, Peoria, Arizona
  - Regeneron Investigational Site, Anaheim, California
  - Regeneron Investigational Site, Beverly Hills, California
  - Regeneron Investigational Site, National City, California
  - Regeneron Investigational Site, Santa Ana, California
  - Regeneron Investigational Site, Milford, Connecticut
  - Regeneron Investigational Site, Stamford, Connecticut
  - Regeneron Investigational Site, Clearwater, Florida
  - Regeneron Investigational Site, Hallandale, Florida
  - Regeneron Investigational Site, St. Petersburg, Florida
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, West Palm Beach, Florida
  - Regeneron Investigational Site, Atlanta, Georgia
  - Regeneron Investigational Site, Sandy Springs, Georgia
  - Regeneron Investigational Site, Overland Park, Kansas
  - Regeneron Investigational Site, Rockville, Maryland
  - Regeneron Investigational Site, Kansas City, Missouri
  - Regeneron Investigational Site, Albuquerque, New Mexico
  - Regeneron Investigational Site, Raleigh, North Carolina
  - Regeneron Investigational Site, Cincinnati, Ohio
  - Regeneron Investigational Site, Duncansville, Pennsylvania
  - Regeneron Investigational Site, Tyrone, Pennsylvania
  - Regeneron Investigational Site, Warwick, Rhode Island
  - Regeneron Investigational Site, Greer, South Carolina
  - Regeneron Investigational Site, Memphis, Tennessee
  - Regeneron Investigational Site, El Paso, Texas
  - Regeneron Investigational Site, San Antonio, Texas
  - Regeneron Invesitgational Site, West Jordan, Utah